CLINICAL TRIAL: NCT07379177
Title: Evaluation of the Pharmacokinetics of Curcumin Capsules in Healthy Human
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kingdomway (Inner Mongolia) Nutritional Food Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: [2026]Ethical Audit No. (001)
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: curcumin
MeSH Terms: interventions — Curcumin; nanocurcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nano Curcumin Capsules (Experimental): Test Group
  Interventions: Dietary Supplement: Nanocurcumin
- Curcumin Capsules (Active Comparator): Reference Group
  Interventions: Dietary Supplement: Curcumin

INTERVENTIONS:
Dietary Supplement: Curcumin — In the first cycle, take 4 capsules of the self-developed product (T, Nano Curcumin Capsules) (125 mg per capsule), in the second cycle take 2 capsules of the control product (R, Curcumin Capsules) (250 mg per capsule), take with 240 mL of water, and the cleansing period is 7 days.
  Arms: Curcumin Capsules
Dietary Supplement: Nanocurcumin — In the first cycle, take 2 capsules (250mg each) of the control product (R, Curcumin Capsules). In the second cycle, take 4 capsules (125mg each) of the self-developed product (T, Nano Curcumin Capsules). Take with 240 mL of water and the cleansing period is 7 days.
  Arms: Nano Curcumin Capsules

SUMMARY:
Main objective:

Through blood drug concentration testing, evaluate the post-meal pharmacokinetic characteristics of the curcumin product compared to similar products, and assess the differences in body exposure between the self-developed product and the control product in healthy trial participants.

Secondary objective:

Observe the safety of the self-developed product and the control product in healthy trial participants.

Study population:

Healthy male individuals or non-pregnant non-lactating females

ELIGIBILITY:
Inclusion Criteria:

1. Both men and women are eligible; women must be non-pregnant and non-lactating.
2. Healthy trial participants aged 18 to 65 years (inclusive of the threshold value).
3. Body Mass Index (BMI) = weight (kg) / height² (m²), with BMI within the range of 18.5 to 30.0 kg/m² (including the threshold value); male trial participants must have a weight of ≥ 50.0 kg, and female trial participants must have a weight of ≥ 45.0 kg.
4. Voluntary participants who have signed the informed consent form; the process of obtaining the informed consent form complies with GCP.
5. Female trial participants agree to use effective non-pharmacological methods for appropriate contraception 2 weeks before the trial diet (for male trial participants, starting from the first trial diet), and within 3 months after the last trial diet, and have no plans for egg donation (male sperm donation).

Exclusion Criteria:

1. Select those who have abnormal and clinically significant findings in physical examination, vital sign examination, blood routine, blood biochemistry, coagulation function, blood pregnancy test (only for females), urine routine, 12-lead electrocardiogram, HBsAg, HCV antibody, HIV antibody, syphilis screening, etc.;
2. Those with a history of serious diseases in cardiovascular, endocrine, digestive, respiratory, urinary, immune system and nervous system, or those who developed the above-mentioned diseases during the screening period, and whose research doctors consider them unsuitable to participate in the clinical trial;
3. Those who are allergic to two or more drugs or foods (including lactose-intolerant individuals); or those who are prone to asthma, rash, urticaria, etc.; or those who have a known history of allergy to curcumin or any excipients;
4. Those with a history of mental illness, drug abuse history, or drug dependence history;
5. Those who have used any prescription drugs, over-the-counter drugs, herbal medicine or health supplements within 14 days before the first trial meal (excluding topical preparations or local drug preparations);
6. Those who have smoked an average of more than 5 cigarettes per day within the previous 3 months;
7. Those who have difficulty in blood collection or cannot tolerate venipuncture blood collection;
8. Those who have a history of heavy drinking (more than 14 units of alcohol per day, 1 unit = 360 mL beer or 45 mL 40% spirituous alcohol or 150 mL wine) or who do not agree to stop consuming alcoholic products during the trial period (from the screening day to the last cycle discharge);
9. Those who have used drugs within the previous 3 months, or those with a positive drug abuse screening result;
10. Those who have consumed excessive tea, coffee or caffeine-containing beverages (more than 8 cups, 1 cup = 250 mL) every day within the previous 3 months;
11. Those who have donated blood or suffered massive blood loss (more than 200 mL) within the previous 3 months;
12. Those who participated in any drug clinical trial and used any clinical trial drugs within the previous 3 months;
13. Those with special dietary requirements and cannot follow the unified diet;
14. Those who have taken special diets or other diets that affect drug absorption, distribution, metabolism, and excretion factors within 7 days before the first trial meal;
15. Those who have had acute diseases during the screening stage or before the allocation of the trial number;
16. Those whose alcohol breath test result is not 0 mg/100 mL within the first cycle;
17. Those who voluntarily withdraw from the trial;
18. Those judged by the researchers to be unsuitable to participate;
19. The number of participants has reached the limit and the screening number of this trial participant is at the rear.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-28 (Estimated); Primary Completion 2026-02-07 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) 0-t | 2 weeks
  plasma concentration-time curve from zero to the time of the last measurable time point t
Peak Plasma Concentration (Cmax) | 2 weeks
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC)0-∞ | 2 weeks
  area under the plasma concentration-time curve from zero to infinity

CONTACTS AND LOCATIONS:
Locations (1):
- No. 55, Zhenhai Road, Xiamen, Fujian, China